CLINICAL TRIAL: NCT03522246
Title: ATHENA (A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study in Ovarian Cancer Patients Evaluating Rucaparib and Nivolumab as Maintenance Treatment Following Response to Front-Line Platinum-Based Chemotherapy)
Brief Title: A Study in Ovarian Cancer Patients Evaluating Rucaparib and Nivolumab as Maintenance Treatment Following Response to Front-Line Platinum-Based Chemotherapy
Acronym: ATHENA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Gynecologic Oncology Group (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO-338-087/GOG-3020/ENGOT-ov45; 2017-004557-17 (EudraCT Number); 2024-516662-11-00 (EU CTIS Number)
Record Dates: First submitted 2018-04-09; First posted 2018-05-11 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal; Fallopian Tube Cancer; Newly Diagnosed; FIGO Stage III-IV; Partial Response; Complete Response
Keywords: PARP inhibitor; PARPi; HRD; ATHENA; homologous recombination; DNA repair; LOH; DNA defect; DNA anomaly; Rucaparib; Nivolumab; PD-1; Immuno-; oncology; Tumor; mutational; burden; BRCA; First-line; Primary Therapy; Primary Treatment
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Pathologic Complete Response; Neoplasms | interventions — rucaparib; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind; only the safety cohort will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (Experimental): Oral rucaparib + intravenous (IV) nivolumab
  Interventions: Drug: Rucaparib; Drug: Nivolumab
- Arm B (Experimental): Oral rucaparib + IV placebo
  Interventions: Drug: Rucaparib; Drug: Placebo IV Infusion
- Arm C (Experimental): Oral placebo + IV nivolumab
  Interventions: Drug: Nivolumab; Drug: Placebo Oral Tablet
- Arm D (Placebo Comparator): Oral placebo + IV placebo
  Interventions: Drug: Placebo Oral Tablet; Drug: Placebo IV Infusion
- Japanese Open-label Safety Cohort (Experimental): Oral rucaparib + IV nivolumab
  Interventions: Drug: Rucaparib; Drug: Nivolumab

INTERVENTIONS:
Drug: Rucaparib — Oral rucaparib will be administered twice daily
  Other Names: Rubraca; CO-338
  Arms: Arm A; Arm B; Japanese Open-label Safety Cohort
Drug: Nivolumab — IV nivolumab will be administered once every 4 weeks
  Other Names: Opdivo; BMS-936558
  Arms: Arm A; Arm C; Japanese Open-label Safety Cohort
Drug: Placebo Oral Tablet — Placebo tablets will be administered twice daily
  Arms: Arm C; Arm D
Drug: Placebo IV Infusion — IV placebo will be administered once every 4 weeks
  Arms: Arm B; Arm D

SUMMARY:
This is a Phase 3, randomized, multinational, double-blind, dual placebo-controlled, 4-arm study evaluating rucaparib and nivolumab as maintenance treatment following response to front-line treatment in newly diagnosed ovarian cancer patients. Response to treatment will be analyzed based on homologous recombination (HR) status of tumor samples.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed advanced (FIGO stage III-IV) epithelial ovarian, fallopian tube, or primary peritoneal cancer.
* Completed cytoreductive surgery, including at least a bilateral salpingo-oophorectomy and partial omentectomy, either prior to chemotherapy (primary surgery) or following neoadjuvant chemotherapy (interval debulking)
* Completed first-line platinum-based chemotherapy and surgery with a response, in the opinion of the Investigator
* Sufficient tumor tissue for planned analysis
* ECOG performance status of 0 or 1
* Patients must be 20 years of age to consent in Japan, Taiwan and South Korea; in all other participating countries patients must be 18 years of age to consent

Exclusion Criteria:

* Pure sarcomas or borderline tumors or mucinous tumors
* Active second malignancy
* Known central nervous system brain metastases
* Any prior treatment for ovarian cancer, other than the first-line platinum regimen
* Evidence of interstitial lung disease or active pneumonitis
* Active, known or suspected autoimmune disease
* Condition requiring active systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1097 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2030-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (238):
- United States (64):
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - John Muir Clinical Research Center, Concord, California
  - UCLA Women's Health Clinical Research Unit, Los Angeles, California
  - Kaiser Permanente Northern California, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Yale University, New Haven, Connecticut
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - MD Anderson Cancer Center-Baptist, Jacksonville, Florida
  - Baptist Health Medical Group Oncology, LLC, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Northside Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Dr. Sudarshan K. Sharma, Ltd - Gynecologic Oncology, Hinsdale, Illinois
  - Ferrell-Duncan Clinic, Springfield, Illinois
  - Community Health Network, Indianapolis, Indiana
  - University of Iowa Hospitals, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Scarborough, Maine
  - SKCCC at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Women's Cancer Care Associates, Albany, New York
  - Broome Oncology, LLC, Johnson City, New York
  - Northwell Health Monter Cancer Center, Lake Success, New York
  - New York University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center - Ohio Health, Columbus, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - LMG Gynecologic Oncology, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Abington Memorial Hospital, Willow Grove, Pennsylvania
  - Avera Gynecologic Oncology, Sioux Falls, South Dakota
  - Texas Oncology - Austin Central, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Memorial Hermann, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - The Woodlands, Gynecologic Oncology, The Woodlands, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Northern Cancer Institute St Leonards, Saint Leonards, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Brian Fricker Oncology Centre, Burnside Hospital, Toorak Gardens, South Australia
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- UZ Leven, Leuven, Belgium
- Canada (13):
  - Alberta Health Services - University of Calgary, Calgary, Alberta
  - Alberta Health Services and The University of Alberta, Edmonton, Alberta
  - BC Cancer - Abbotsford, Abbotsford, British Columbia
  - BC Cancer - Kelowna, Kelowna, British Columbia
  - BC Cancer - Surrey, Surrey, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nsha-Qeii Hsc, Halifax, Nova Scotia
  - Juravinski Cancer Center, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Centre Hospitalier de l'Université de Montreal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Centre Integre Universitaire de sante et de service sociaux de l'Estri-Centre hospitalier univeritaire de Sherbrooke, Sherbrooke, Quebec
- Czechia (3):
  - Masaryk Memorial Cancer Institute, Brno
  - Department of Gynecology and Obstetrics, Oncogynecological center U hiversity Hospital Kralovske Vinohrady, Prague
  - KOC KNTB a.s. Zlfn, Hvalfckovo nabrezf 600, 76001, Zlín
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Odense University Hospital, Odense
- Kuopio University Hospital, Kuopio, Finland
- Germany (5):
  - Klinik für Frauenheilkunde und Geburtshilfe, Dessau
  - Universitaetsklinikum Duesseldorf / Klinik fur Frauenheilkunde & Geburtshilfe, Düsseldorf
  - Universitatsklinikum National Centrum for Tumor Disease (NCT), Heidelberg
  - Universitätslinikum Mannheim, Frauenklinik, Mannheim
  - Kliniken Suedostbayern AG, Klinikum Traunstein, Traunstein
- Greece (5):
  - Attikon General University Hospital, Chaïdári, Athens
  - University Hospital Attikon, Chaïdári, Athens
  - Alexandra Hospital, Athens
  - General Hospital of Patras, Pátrai
  - Euromedica General Clinic, B' Oncology Clinic, Thessaloniki
- Ireland (4):
  - Cork University Hospital, Cork
  - Bon Secours Hospital, Cork
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford
- Israel (6):
  - Shaare Zedek Medical Oncology, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Sheba Medical Center, Ramat Gan
  - Ziv Medical Center, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Centro di Riferimento Oncologico, CRO-IRCCS, Aviano
  - Candiolo Cancer Institute - IRCCS, Candiolo
  - Arnas Garibaldi, Catania
  - University G, D'Annunuzio-Chieti, Chieti
  - IRCCS Instituto Nazionale Tumori, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Umberto I, Roma
  - Policlinico Agostino Gemelli, Roma
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma
  - Ospedale San Bortolo, Vicenza
- Japan (20):
  - University of Tsukuba Hospital, Tsukuba, Amakubo
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Yokohama City University Hospital, Yokohama, Fukuura
  - Gunma University Hospital, Maebashi, Gunma
  - Gunma Prefectural Cancer Center, Ota-shi, Gunma
  - Hiroshima City Hiroshima Citizens Hospital, Naka, Hiroshima
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Iwate Medical University, Morioka, Iwate
  - Nippon Medical School Musashikosugi Hospital, Kawasaki-shi, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Defense Medical College Hospital, Tokorozawa, Namiki
  - Osaka International Cancer Institute, Chuo, Osaka
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Keio University Hospital, Shinjuku-Ku, Shinanomachi
  - The Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - Saitama Cancer Center, Saitama
  - Kagawa Prefectural Central Hospital, Takamatsu
  - National Cancer Center Hospital, Tokyo
- New Zealand (5):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North
  - Tauranga Hospital, Tauranga
- Poland (7):
  - Chair & department of Obsterics, Gynaecology and Oncology (previous site), Warsaw, Kondratowicza
  - Bialostockie Centrum Onkologii Oddzial Onkologii Ginekologicznej, Bialystok
  - University Hospital of Bialystok, Bialystok
  - Szpitale Pomorskie sp zoo, Gdynia
  - Medical University of Lublin, Lublin
  - Wielkopolskie Centrum Onkologii, Poznan
  - Pomeranian Medical University, Szczecin
- Romania (11):
  - Spitalul Clinic Municipal "Dr. Gavril Curteanu", Oradea, Jud. Bihor
  - S.C. Medisprof S.R.L., Cluj-Napoca, Jud. Cluj
  - Oncopremium Team, Baia Mare
  - SC Quantum Medical Center SRL, Bucharest
  - Instiute of Oncology - Medical Oncology, Cluj-Napoca
  - Centrul de Oncologie Sf.Nectarie, Craiova
  - S.C Oncolab S.R.L, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spital Municipal Ploiesti, Ploieşti
  - Spitalul Judetean de Urgenta "Sfantul Ioan cel Nou" Suceava, Suceava
  - ONCOMED Timisoara, Timișoara
- Russia (11):
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - BHI of Omsk Region Clinical Oncology Dispensary, Omsk
  - Orenburg Regional Clinical Oncological Dispensary, Orenburg
  - SBHI Saint Petersburg Research Center specialized types of medical care (Oncology), Pesochnyy
  - SBHI SR Pyatigorsk Interdistrict Oncology Dispensary, Pyatigorsk
  - Limited Liability Company MedPomosch, Saint Petersburg
  - FSBEI HE I.P. Pavlov SPbSMU MoH Russia, Saint Petersburg
  - Saint-Petersburg State Budget Institution of Healthcare City Clinical Oncology Dispensary, Saint Petersburg
  - 1st Medical University, Saint Petersburg
  - Federa; State Budgetary Educational Institution of Higher Education National Research Ogarev Mordovia State University, Saransk
  - State Medical Institution "Oncology Center #2" under the Krasnodar Region Healthcare Department, Sochi
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Center Singapore, Singapore
- South Korea (13):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Seoul
  - SoonChunHyang University Cheonan Hospital, Cheonan
  - Korea Cancer Center Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (10):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Consorcio Hospitalario Provincial Castellon, Castillón
  - Hospital Virgen de la Arrixaca, El Palmar
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Nuestra Señora de Valme, Seville
- Sweden (3):
  - Onkologiska Kliniken, Linköping
  - Onkologiska Kliniken, Lund
  - Karolinska Universitetssjukhuset, Stockholm
- Taiwan (13):
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Chi Mei Hospital, Liouying (CMHLY), Tainan
  - Chi Mei Medical Center (CMMC), Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Medical Foundation- Linkou Branch, Taoyuan District
- Turkey (Türkiye) (5):
  - Dr. Abdurrahman Yurtaslan Ankara Women's Health Education and Research Hospital, Ankara
  - Istanbul University-cerrahpasa, Cerrahpasa School of Medicine, Istanbul
  - Koc University School of Medicine, Koc University Hospital, Istanbul
  - Celal Bayar University Faculty of Medicine, Manisa
  - Baskent University Hospital, Yüreğir
- United Kingdom (17):
  - East Kent Hospitals University NHS Foundation trust Medical Oncology, Canterbury, Kent
  - Northampton General Hospital, Cliftonville, Northampton
  - Royal Sussex County Hospital, Brighton
  - Bristol Cancer Institute Medical Oncology, Bristol
  - Addenbrookes Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster
  - St. James University Hospital, Leeds
  - Barts and the London NHS Trust, London
  - University of College London Hospital, London
  - Guy's & St Thomas' NHS Foundation Trust (Guy's Cancer Centre), London
  - The Royal Marsden NHS Foundation Trust, London
  - Imperial College London, London
  - The James Cook University Hospital, Middlesbrough
  - Poole Hospital NHS Foundation Trust, Poole
  - South West Wales Cancer Centre - Singleton Hospital, Swansea
  - Musgrove Park Hospital, Taunton

REFERENCES:
- [Derived] Monk BJ, Parkinson C, Lim MC, O'Malley DM, Oaknin A, Wilson MK, Coleman RL, Lorusso D, Bessette P, Ghamande S, Christopoulou A, Provencher D, Prendergast E, Demirkiran F, Mikheeva O, Yeku O, Chudecka-Glaz A, Schenker M, Littell RD, Safra T, Chou HH, Morgan MA, Drochytek V, Barlin JN, Van Gorp T, Ueland F, Lindahl G, Anderson C, Collins DC, Moore K, Marme F, Westin SN, McNeish IA, Shih D, Lin KK, Goble S, Hume S, Fujiwara K, Kristeleit RS. A Randomized, Phase III Trial to Evaluate Rucaparib Monotherapy as Maintenance Treatment in Patients With Newly Diagnosed Ovarian Cancer (ATHENA-MONO/GOG-3020/ENGOT-ov45). J Clin Oncol. 2022 Dec 1;40(34):3952-3964. doi: 10.1200/JCO.22.01003. Epub 2022 Jun 6. PMID 35658487
- [Derived] Monk BJ, Coleman RL, Fujiwara K, Wilson MK, Oza AM, Oaknin A, O'Malley DM, Lorusso D, Westin SN, Safra T, Herzog TJ, Marme F, N Eskander R, Lin KK, Shih D, Goble S, Grechko N, Hume S, Maloney L, McNeish IA, Kristeleit RS. ATHENA (GOG-3020/ENGOT-ov45): a randomized, phase III trial to evaluate rucaparib as monotherapy (ATHENA-MONO) and rucaparib in combination with nivolumab (ATHENA-COMBO) as maintenance treatment following frontline platinum-based chemotherapy in ovarian cancer. Int J Gynecol Cancer. 2021 Dec;31(12):1589-1594. doi: 10.1136/ijgc-2021-002933. Epub 2021 Sep 30. PMID 34593565

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment is complete and the study is ongoing. Data are presented here for the primary endpoint analysis.
Groups:
- Arm A: Rucaparib + Nivolumab: Participants received oral rucaparib tablets twice daily and nivolumab intravenous (IV) infusion once every 4 weeks.
- Arm B: Rucaparib + Placebo: Participants received oral rucaparib tablets twice daily and placebo IV infusion once every 4 weeks.
- Arm C: Placebo + Nivolumab: Participants received oral placebo tablets twice daily and nivolumab IV infusion once every 4 weeks.
- Arm D: Placebo + Placebo: Participants received oral placebo tablets twice daily and placebo IV infusion once every 4 weeks.
- Japanese Open-label Safety Cohort: Rucaparib + Nivolumab: Participants received oral rucaparib tablets twice daily and nivolumab IV infusion once every 4 weeks.
Period: Overall Study
Arm/Group | Arm A: Rucaparib + Nivolumab | Arm B: Rucaparib + Placebo | Arm C: Placebo + Nivolumab | Arm D: Placebo + Placebo | Japanese Open-label Safety Cohort: Rucaparib + Nivolumab
Started | 436 | 427 | 108 | 111 | 15
Received at Least 1 Dose of Study Drug | 433 | 425 | 108 | 110 | 15
Safety Population (The Safety Population consisted of all participants who received at least 1 dose of protocol-specified treatment (oral and/or IV study drug). For safety analyses, data were presented separately for all treatment arms according to actual treatment given, such that participants randomized to either treatment group containing IV nivolumab (ie, Arms A or C) who never received nivolumab were then analyzed in the analogous treatment group that contained IV placebo (ie, Arms B or D, respectively).) | 410 | 448 | 107 | 111 | 15
Completed (Study completion was defined as completion due to death, loss to follow-up, COVID-19, withdrawal of consent, or study closure.) | 252 | 233 | 62 | 66 | 15
Not Completed | 184 | 194 | 46 | 45 | 0
Not completed — Ongoing in Long-Term Follow-up (Alive) | 184 | 194 | 46 | 45 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Arm A: Rucaparib + Nivolumab; Japanese Open-label Safety Cohort: Rucaparib + Nivolumab: Participants received oral rucaparib tablets twice daily and nivolumab IV infusion once every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm A: Rucaparib + Nivolumab | Arm B: Rucaparib + Placebo | Arm C: Placebo + Nivolumab | Arm D: Placebo + Placebo | Japanese Open-label Safety Cohort: Rucaparib + Nivolumab | Total
Number analyzed (Participants) | 436 | 427 | 108 | 111 | 15 | 1097
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 281 | 270 | 72 | 68 | 13 | 704
  >=65 years | 155 | 157 | 36 | 43 | 2 | 393
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 436 | 427 | 108 | 111 | 15 | 1097
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 1 | 1 | 0 | 34
  Not Hispanic or Latino | 405 | 397 | 102 | 107 | 14 | 1025
  Unknown or Not Reported | 16 | 13 | 5 | 3 | 1 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 1 | 0 | 4
  Asian | 81 | 80 | 22 | 16 | 15 | 214
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 0 | 1 | 0 | 5
  Black or African American | 8 | 5 | 1 | 3 | 0 | 17
  White | 325 | 328 | 83 | 87 | 0 | 823
  More than one race | 0 | 2 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 19 | 8 | 2 | 2 | 0 | 31

OUTCOME MEASURES:

1. Primary Outcome: Monotherapy Arm B and Arm D: Investigator Assessed Progression-free Survival (PFS)
Description: PFS by investigator was defined as the time from randomization to disease progression, according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as assessed by the investigator, or death due to any cause, whichever occurred first.
  Progressive disease was defined as a 20% increase in the sum of the longest diameter of measurable lesions, an unequivocal increase in existing non-measurable lesion(s), or the appearance of unequivocal new lesion(s).
Time Frame: From randomization until disease progression (up to the primary data analysis at approximately 39 months)
Population: The homologous recombination deficiency (HRD) population consisted of all randomized participants with either a tumor tissue alteration in breast cancer genes (BRCA)1 or BRCA2 (tBRCA) or non-tBRCA high loss of heterozygosity (LOHhigh). Presented here are data for the monotherapy comparison arms (Arm B and Arm D).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 185 | 49
months | 28.7 [23.0 to NA] — Not reached due to insufficient number of events | 11.3 [9.1 to 22.1]
Statistical Analysis 1: Comparison: Arm B: Rucaparib + Placebo vs Arm D: Placebo + Placebo; Test type: Superiority — Rucaparib vs Placebo; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.31 to 0.72] — The stratified cox proportional hazard model is adjusted for the randomization strata of HRD classification and timing of surgery

2. Primary Outcome: Monotherapy Arm B and Arm D: Investigator Assessed PFS
Description: PFS by investigator was defined as the time from randomization to disease progression, according to RECIST v1.1 as assessed by the investigator, or death due to any cause, whichever occurred first.
  Progressive disease was defined as a 20% increase in the sum of the longest diameter of measurable lesions, an unequivocal increase in existing non-measurable lesion(s), or the appearance of unequivocal new lesion(s).
Time Frame: From randomization until disease progression (up to the primary data analysis at approximately 39 months)
Population: The ITT population included all randomized participants. Presented here are data for the monotherapy comparison arms (Arm B and Arm D).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 427 | 111
months | 20.2 [15.2 to 24.7] | 9.2 [8.3 to 12.2]
Statistical Analysis 1: Comparison: Arm B: Rucaparib + Placebo vs Arm D: Placebo + Placebo; Test type: Superiority — Rucaparib vs Placebo; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.40 to 0.68] — The stratified cox proportional hazard model is adjusted for the randomization strata of HRD classification, disease status post-chemotherapy, and timing of surgery

3. Primary Outcome: Combination Therapy Arm A and Arm B: Investigator Assessed PFS
Description: as for outcome 2
Time Frame: From randomization until disease progression (up to the combination therapy interim analysis at approximately 66 months)
Population: The ITT population included all randomized participants. Presented here are data from combination comparison arms (Arm A and Arm B).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Rucaparib + Nivolumab | Arm B: Rucaparib + Placebo
Number analyzed (Participants) | 436 | 427
months | 15.0 [12.1 to 17.4] | 20.2 [15.6 to 24.0]
Statistical Analysis 1: Comparison: Arm A: Rucaparib + Nivolumab vs Arm B: Rucaparib + Placebo; Test type: Superiority — Rucaparib + Nivolumab vs Rucaparib + Placebo; p = 0.0038, Log Rank; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [1.08 to 1.53] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Monotherapy Arm B and Arm D: Blinded Independent Central Review (BICR) PFS
Description: PFS was assessed by BICR per RECIST v1.1 as the time from randomization to disease progression, or death due to any cause, whichever occurred first.
  Progressive disease was defined as a 20% increase in the sum of the longest diameter of measurable lesions, an unequivocal increase in existing non-measurable lesion(s), or the appearance of unequivocal new lesion(s).
Time Frame: From randomization until disease progression (up to the primary data analysis at approximately 39 months)
Population: The HRD population consisted of all randomized participants with either tBRCA or non-tBRCA LOHhigh. Presented here are data from the monotherapy comparison arms (Arm B and Arm D).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 185 | 49
months | NA [28.7 to NA] — Not reached due to insufficient number of events | 9.9 [6.5 to NA] — Not reached due to insufficient number of events

5. Secondary Outcome: Monotherapy Arm B and Arm D: BICR PFS
Description: as for outcome 4
Time Frame: From randomization until disease progression (up to the primary data analysis at approximately 39 months)
Population: The ITT population included all randomized participants. Presented here are data from the monotherapy comparison arms (Arm B and Arm D).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 427 | 111
months | 25.9 [16.8 to NA] — Not reached due to insufficient number of events | 9.1 [6.4 to 9.7]

6. Secondary Outcome: Combination Therapy Arm A and Arm B: BICR PFS
Description: as for outcome 4
Time Frame: as for outcome 3
Population: BICR was included as a supportive secondary endpoint in the event that the Investigator-assessed PFS result was positive. In the ATHENA-COMBO statistical analysis plan it was specified that the BICR analysis would only be performed if the primary endpoint of Investigator-assessed PFS was statistically significant. Given that the result was negative and not statistically significant, the analysis of BICR was not performed, thus that data is not available and cannot be provided.
Arm/Group | Arm A: Rucaparib + Nivolumab | Arm B: Rucaparib + Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Monotherapy Arm B and Arm D: Overall Survival (OS)
Description: OS was defined as the number of days (measured in months) from the date of randomization to the date of death due to any cause.
Time Frame: From randomization until death due to any cause (up to the primary data analysis at approximately 36 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 185 | 49
months | NA [NA to NA] — Not reached due to insufficient number of events. | NA [NA to NA] — Not reached due to insufficient number of events.

8. Secondary Outcome: Monotherapy Arm B and Arm D: OS
Description: as for outcome 7
Time Frame: From randomization until death due to any cause (up to the primary data analysis at approximately 40 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 427 | 111
months | 38.8 [38.8 to NA] — Not reached due to insufficient number of events. | NA [31.4 to NA] — Not reached due to insufficient number of events.

9. Secondary Outcome: Combination Therapy Arm A and Arm B: OS
Description: as for outcome 7
Time Frame: From randomization until death due to any cause (up to the combination therapy interim analysis at approximately 72 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Rucaparib + Nivolumab | Arm B: Rucaparib + Placebo
Number analyzed (Participants) | 436 | 427
months | 49.4 [43.9 to 55.3] | 58.0 [46.7 to NA] — Not reached due to insufficient number of events

10. Secondary Outcome: Monotherapy Arm B and Arm D: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed Complete Response (CR) or Partial Response (PR) as assessed by the Investigator per RECIST 1.1.
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization until disease progression (up to the primary data analysis at approximately 39 months)
Population: The HRD population consisted of all randomized participants with either tBRCA or non-tBRCA LOHhigh. Presented here are data from the monotherapy comparison arms (Arm B and Arm D). Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 17 | 5
percentage of participants | 58.8 [32.9 to 81.6] | 20.0 [0.5 to 71.6]

11. Secondary Outcome: Monotherapy Arm B and Arm D: ORR
Description: ORR was defined as the percentage of participants with CR or PR as assessed by the Investigator per RECIST 1.1.
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization until disease progression (up to the primary data analysis at approximately 39 months)
Population: The ITT population included all randomized participants. Presented here are data from the monotherapy comparison arms (Arm B and Arm D). Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 41 | 11
percentage of participants | 48.8 [32.9 to 64.9] | 9.1 [0.2 to 41.3]

12. Secondary Outcome: Combination Therapy Arm A and Arm B: ORR
Description: as for outcome 11
Time Frame: as for outcome 3
Population: The ITT population included all randomized participants. Presented here are data from combination comparison arms (Arm A and Arm B). Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Rucaparib + Nivolumab | Arm B: Rucaparib + Placebo
Number analyzed (Participants) | 39 | 41
percentage of participants | 25.6 [13.0 to 42.1] | 48.8 [32.9 to 64.9]

13. Secondary Outcome: Monotherapy Arm B and Arm D: Duration of Response (DOR)
Description: DOR was assessed by the investigator and defined as the interval from the first documentation of objective response (CR or PR per RECIST v1.1) to the earlier of the first documentation of progressive disease (PD) or death from any cause.
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  PD: 20% increase in the sum of the longest diameter of measurable lesions, an unequivocal increase in existing non-measurable lesion(s), or the appearance of unequivocal new lesion(s).
Time Frame: From first confirmed response until disease progression (up to the primary data analysis at approximately 30 months)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 10 | 1
months | 16.7 [5.7 to NA] — Not reached due to insufficient number of events | 5.5 [NA to NA] — Not reached due to insufficient number of events

14. Secondary Outcome: Monotherapy Arm B and Arm D: DOR
Description: DOR was assessed by the investigator and defined as the interval from the first documentation of objective response (CR or PR per RECIST v1.1) to the earlier of the first documentation of PD or death from any cause.
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  PD: 20% increase in the sum of the longest diameter of measurable lesions, an unequivocal increase in existing non-measurable lesion(s), or the appearance of unequivocal new lesion(s).
Time Frame: From first confirmed response until disease progression (up to the primary data analysis at approximately 33 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Arm B: Rucaparib + Placebo | Arm D: Placebo + Placebo
Number analyzed (Participants) | 20 | 1
months | 22.1 [8.4 to NA] — Not reached due to insufficient number of events | 5.5 [NA to NA] — Not reached due to insufficient number of events

15. Secondary Outcome: Combination Therapy Arm A and Arm B: DOR
Description: as for outcome 14
Time Frame: From first confirmed response until disease progression (up to the combination therapy interim analysis at approximately 60 months)
Population: The ITT population included all randomized participants. Presented here are data from the combination comparison arms (Arm A and Arm B). Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Arm A: Rucaparib + Nivolumab | Arm B: Rucaparib + Placebo
Number analyzed (Participants) | 10 | 20
months | 13.7 [5.6 to NA] — Not reached due to insufficient number of events | 27.7 [8.4 to NA] — Not reached due to insufficient number of events

ADVERSE EVENTS:
Time Frame: Up to approximately 5 years
Description: The Safety Population consisted of all participants who received at least 1 dose of protocol-specified treatment (oral and/or IV study drug). For safety analyses, data were presented separately for all treatment arms according to actual treatment given, such that participants randomized to either treatment group containing IV nivolumab (ie, Arms A or C) who never received nivolumab were then analyzed in the analogous treatment group that contained IV placebo (ie, Arms B or D, respectively).
Arm/Group | Arm A: Rucaparib + Nivolumab | Arm B: Rucaparib + Placebo | Arm C: Placebo + Nivolumab | Arm D: Placebo + Placebo | Japanese Open-label Safety Cohort: Rucaparib + Nivolumab
All-Cause Mortality (participants affected / at risk) | 12/410 | 20/448 | 4/107 | 2/111 | 0/15
Serious Adverse Events (participants affected / at risk) | 154/410 | 117/448 | 18/107 | 13/111 | 4/15
Other Adverse Events (participants affected / at risk) | 406/410 | 433/448 | 99/107 | 103/111 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Rucaparib + Nivolumab (N=410) | Arm B: Rucaparib + Placebo (N=448) | Arm C: Placebo + Nivolumab (N=107) | Arm D: Placebo + Placebo (N=111) | Japanese Open-label Safety Cohort: Rucaparib + Nivolumab (N=15)
Anaemia (Blood and lymphatic system disorders) | 23 (35) | 18 (20) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 30 (37) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 10 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vogt-Koyanagi-Harada disease (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 11 (14) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (10) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brucellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected lymphocele (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (7) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Product administration error (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma prolapse (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 16 (16) | 3 (3) | 1 (1) | 0 (0)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic neurological syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Rucaparib + Nivolumab (N=410) | Arm B: Rucaparib + Placebo (N=448) | Arm C: Placebo + Nivolumab (N=107) | Arm D: Placebo + Placebo (N=111) | Japanese Open-label Safety Cohort: Rucaparib + Nivolumab (N=15)
Anaemia (Blood and lymphatic system disorders) | 198 (789) | 198 (778) | 10 (23) | 11 (23) | 12 (49)
Leukopenia (Blood and lymphatic system disorders) | 40 (118) | 18 (69) | 1 (1) | 3 (8) | 4 (7)
Lymphopenia (Blood and lymphatic system disorders) | 12 (21) | 9 (20) | 0 (0) | 1 (1) | 2 (6)
Neutropenia (Blood and lymphatic system disorders) | 89 (300) | 65 (216) | 5 (5) | 8 (18) | 6 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 78 (198) | 51 (126) | 2 (2) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 8 (9) | 6 (6) | 2 (2) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 26 (33) | 3 (3) | 11 (12) | 3 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 40 (57) | 12 (14) | 14 (19) | 5 (7) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 15 (24) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Vitreous floaters (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 33 (40) | 44 (56) | 3 (3) | 15 (17) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 91 (139) | 109 (146) | 15 (21) | 32 (45) | 4 (8)
Abdominal pain upper (Gastrointestinal disorders) | 35 (46) | 42 (55) | 5 (5) | 9 (15) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 100 (137) | 85 (125) | 11 (12) | 17 (20) | 1 (1)
Dental caries (Gastrointestinal disorders) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 113 (217) | 107 (181) | 20 (34) | 25 (41) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 20 (22) | 16 (16) | 7 (11) | 5 (7) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 30 (38) | 44 (55) | 5 (5) | 9 (11) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (18) | 21 (23) | 5 (6) | 4 (4) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 7 (7) | 7 (7) | 2 (3) | 2 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 234 (458) | 254 (457) | 27 (32) | 34 (52) | 10 (24)
Stomatitis (Gastrointestinal disorders) | 38 (59) | 34 (72) | 7 (10) | 4 (6) | 4 (8)
Vomiting (Gastrointestinal disorders) | 128 (226) | 107 (187) | 11 (16) | 14 (17) | 4 (6)
Asthenia (General disorders) | 56 (117) | 62 (114) | 7 (11) | 12 (17) | 0 (0)
Fatigue (General disorders) | 186 (384) | 189 (344) | 24 (36) | 34 (56) | 5 (13)
Malaise (General disorders) | 15 (23) | 13 (24) | 2 (4) | 1 (1) | 3 (7)
Non-cardiac chest pain (General disorders) | 5 (6) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Oedema (General disorders) | 10 (11) | 5 (5) | 4 (4) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 32 (45) | 34 (45) | 4 (4) | 13 (15) | 1 (1)
Pyrexia (General disorders) | 65 (97) | 41 (51) | 9 (9) | 6 (9) | 3 (4)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 30 (34) | 27 (29) | 3 (3) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 7 (9) | 12 (13) | 2 (2) | 5 (8) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (3)
Influenza (Infections and infestations) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 16 (21) | 22 (36) | 2 (2) | 2 (2) | 4 (4)
Papilloma viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 2 (3) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 33 (41) | 24 (30) | 8 (9) | 2 (2) | 1 (4)
Urinary tract infection (Infections and infestations) | 52 (80) | 41 (53) | 12 (20) | 12 (19) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 212 (614) | 178 (464) | 17 (28) | 8 (16) | 12 (57)
Amylase increased (Investigations) | 2 (4) | 0 (0) | 1 (3) | 2 (3) | 1 (5)
Aspartate aminotransferase increased (Investigations) | 197 (452) | 161 (341) | 15 (26) | 9 (13) | 14 (39)
Blood alkaline phosphatase increased (Investigations) | 41 (69) | 42 (56) | 2 (3) | 2 (3) | 4 (12)
Blood bilirubin increased (Investigations) | 31 (80) | 19 (40) | 0 (0) | 2 (6) | 1 (3)
Blood cholesterol increased (Investigations) | 30 (48) | 27 (69) | 5 (12) | 3 (7) | 0 (0)
Blood creatinine increased (Investigations) | 66 (162) | 52 (108) | 7 (8) | 6 (11) | 4 (9)
Gamma-glutamyltransferase increased (Investigations) | 9 (14) | 9 (15) | 1 (1) | 0 (0) | 2 (3)
Lymphocyte count decreased (Investigations) | 18 (33) | 12 (26) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 69 (309) | 61 (223) | 6 (15) | 1 (2) | 6 (13)
Platelet count decreased (Investigations) | 65 (240) | 59 (185) | 2 (7) | 0 (0) | 9 (64)
White blood cell count decreased (Investigations) | 58 (217) | 40 (135) | 2 (2) | 3 (5) | 7 (29)
Decreased appetite (Metabolism and nutrition disorders) | 80 (126) | 80 (111) | 7 (13) | 18 (20) | 1 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (3) | 0 (0) | 1 (1) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 14 (28) | 26 (52) | 5 (5) | 7 (10) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 19 (28) | 21 (29) | 1 (1) | 7 (12) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 30 (39) | 23 (34) | 2 (2) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 25 (47) | 32 (52) | 4 (10) | 2 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 19 (34) | 14 (36) | 1 (2) | 7 (9) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 99 (162) | 92 (142) | 24 (42) | 25 (36) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 6 (8) | 10 (11) | 1 (2) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 53 (70) | 45 (62) | 11 (11) | 15 (25) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (11) | 0 (0) | 6 (6) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 (22) | 13 (17) | 3 (4) | 8 (13) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 37 (59) | 54 (76) | 3 (5) | 10 (14) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (38) | 40 (55) | 4 (4) | 8 (16) | 1 (2)
Disturbance in attention (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 65 (82) | 59 (81) | 12 (13) | 11 (14) | 1 (1)
Dysgeusia (Nervous system disorders) | 81 (100) | 91 (125) | 7 (8) | 6 (8) | 8 (14)
Headache (Nervous system disorders) | 78 (127) | 88 (151) | 9 (10) | 18 (35) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 9 (11) | 11 (11) | 2 (2) | 2 (2) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 24 (35) | 37 (45) | 8 (14) | 7 (9) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Taste disorder (Nervous system disorders) | 21 (25) | 24 (24) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 25 (28) | 20 (24) | 2 (2) | 3 (4) | 1 (1)
Depression (Psychiatric disorders) | 18 (21) | 18 (20) | 6 (6) | 2 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 56 (63) | 62 (84) | 8 (9) | 8 (9) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 55 (75) | 56 (75) | 6 (6) | 11 (15) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 67 (106) | 51 (78) | 13 (14) | 13 (16) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 13 (19) | 4 (5) | 4 (5) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (10) | 14 (14) | 1 (2) | 3 (3) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (7) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 22 (31) | 23 (31) | 5 (5) | 2 (2) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 26 (40) | 31 (35) | 1 (1) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 76 (119) | 71 (106) | 8 (8) | 12 (13) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 72 (121) | 65 (95) | 17 (32) | 8 (11) | 4 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 37 (74) | 7 (12) | 2 (5) | 4 (6) | 2 (3)
Hot flush (Vascular disorders) | 15 (17) | 32 (38) | 2 (2) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 26 (39) | 26 (46) | 4 (12) | 8 (15) | 0 (0)
Lymphoedema (Vascular disorders) | 2 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT03522246/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03522246/SAP_001.pdf